CLINICAL TRIAL: NCT05335746
Title: Chorioretinal Changes in Vitiligo Patients on Therapy
Brief Title: Ocular Changes in Vitiligo Patients on Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Abdelshafy, Clinical professor, Benha University
Other Study IDs: Rc 6-2022
Record Dates: First submitted 2022-03-28; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Vitiligo; Chorioretinopathy; Chorioretinitis
Keywords: Vitiligo; Chorioretinitis
MeSH Terms: conditions — Vitiligo; Chorioretinitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vitiligo patients on therapy: Patients diagnosed as vitiligo and on systemic and local therapy.
  Interventions: Diagnostic Test: Optical coherence tomography angiography (OCT-A)
- Control group: Normal subjects recruited from ophthalmology clinic and visit the clinic for regular check-up.
  Interventions: Diagnostic Test: Optical coherence tomography angiography (OCT-A)

INTERVENTIONS:
Diagnostic Test: Optical coherence tomography angiography (OCT-A) — Optical coherence tomography angiography scanning will be done for all subjects in the study.
  Other Names: OCT-A

SUMMARY:
Vitiligo patients on systemic and local therapy may have some ocular adverse effects associated with the disease and its therapy.

DETAILED DESCRIPTION:
Chorioretinal changes associated with vitiligo therapy could address patients visual acuity and life style. Early detection of these changes can help these patients to evade such adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* vitiligo patients on systemic and local therapy that regularly visit dermatology clinic at banha university.
* normal subjects seeking regular ophthalmic examination at ophthalmology clinic at banha university.

Exclusion Criteria:

* patients with known chronic retinal diseases that may alter OCT-A parameters as age related macular degeneration and diabetic retinopathies.
* patients that refuse to participate in this study.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Dermatology and ophthalmology clinics at banha university.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of vessel density (VD) in superficial and deep retinal layer. | Immediately after OCT-A for each eye and at one month of follow-up.
  Percentage (%) of superficial and deep vessel density changes in both groups measured by OCT-A software to asses retinal ischemia.

SECONDARY OUTCOMES:
Foveal avascular zone (FAZ) in millimeter (mm). | Immediately after OCT-A for each eye and at one month of follow-up.
  Foveal avascular zone measurement in both groups in mm measured by OCT-A software.

OTHER OUTCOMES:
Changes in visual acuity | Immediately after OCT-A for each eye and at one month of follow-up.
  Visual acuity measurements in decimal form
Changes in choroidal thickness | Immediately after OCT-A for each eye and at one month of follow-up.
  Choroidal thickness in mm.

CONTACTS AND LOCATIONS:
Overall Officials: Amal A Yousif, MD, Principal Investigator — Benha University
Locations (1):
- Benha University, Banhā, QA, Egypt